CLINICAL TRIAL: NCT05885282
Title: Investigation of the Effects of Local Vibration Applied to Different Regions and Spinal Stabilization Exercises on Postural Control in Patients with Ataxic Multiple Sclerosis
Brief Title: Investigation of the Effects of Local Vibration Applied to Different Regions and Spinal Stabilization Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Local Vibration Application
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis; Ataxia
Keywords: Multiple Sclerosis; ataxia; spinal stabilization; local vibration; postural control
MeSH Terms: conditions — Multiple Sclerosis; Ataxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Exercise Group (Active Comparator): Lumbar spinal stabilization exercises will be given. Lumbar spinal stabilization exercises; diaphragmatic breathing, and contraction of the transversus abdominis and multifidus muscles will be taught in the supine position. Activation of these muscles will be studied in different positions (prone, crawling, sitting, and sitting on different surfaces). The focus will be on increasing kinesthetic awareness. It will be desirable to ensure and maintain the activation of these muscles during subsequent exercises. Exercises will be continued according to the patient's functional status and individual needs. Advancement of exercises; extremity movements on dynamic surfaces, narrowing of support surfaces, reciprocal movements, increasing the number of resistance and repetitions. The duration of a session will be 40 minutes.
  Interventions: Other: Control Exercise
- Paraspinal Vibration Group (Active Comparator): In addition to lumbar spinal stabilization exercises, LV will be applied to the cervical and lumbar paraspinal muscles. Spinal stabilization exercises will be as in the control group. The duration of a session will be 50 minutes, with spinal stabilization exercises 40 minutes and LV 10 minutes.LV will be applied before the exercises. LV will be applied to the cervical paraspinal muscles for a total of 5 minutes (2.5 minutes on the right side, 2.5 minutes on the left side) while the patients are in a sitting position. LV will be applied to the lumbar paraspinal muscles for a total of 5 minutes (2.5 minutes on the right side, 2.5 minutes on the left side) while the patients are lying in the prone position. LV application will be made with Vibrasens © device and vibration frequency 80 Hz amplitude 1 mm will be selected.
  Interventions: Device: paraspinal vibration
- Gastrosoleus Muscle Complex Vibration Group (Active Comparator): In addition to lumbar spinal stabilization exercises, LV will be applied to the gastrosoleus muscle complex. Spinal stabilization exercises will be as in the other 2 groups. The duration of a session will be 50 minutes, with spinal stabilization exercises 40 minutes and LV 10 minutes.LV application will be applied sequentially, bilaterally, to the gastrosoleus complex. LV will be applied before the exercises. LV will be applied for a total of 10 minutes (5 minutes each on the right and left) while the patients are lying in the prone position. LV application will be made with Vibrasens © device and vibration frequency 80 Hz amplitude 1 mm will be selected.
  Interventions: Device: gastrosoleus muscle complex vibration

INTERVENTIONS:
Device: paraspinal vibration — In addition to lumbar spinal stabilization exercises, LV will be applied to the cervical and lumbar paraspinal muscles. Spinal stabilization exercises will be as in the control group. The duration of a session will be 50 minutes, with spinal stabilization exercises 40 minutes and LV 10 minutes.LV will be applied before the exercises. LV will be applied to the cervical paraspinal muscles for a total of 5 minutes (2.5 minutes on the right side, 2.5 minutes on the left side) while the patients are in a sitting position. LV will be applied to the lumbar paraspinal muscles for a total of 5 minutes (2.5 minutes on the right side, 2.5 minutes on the left side) while the patients are lying in the prone position. LV application will be made with Vibrasens © device and vibration frequency 80 Hz amplitude 1 mm will be selected.
  Arms: Paraspinal Vibration Group
Device: gastrosoleus muscle complex vibration — In addition to lumbar spinal stabilization exercises, LV will be applied to the gastrosoleus muscle complex. LV application will be applied sequentially, bilaterally, to the gastrosoleus complex. LV will be applied before the exercises. LV will be applied for a total of 10 minutes (5 minutes each on the right and left) while the patients are lying in the prone position. LV application will be made with Vibrasens © device and vibration frequency 80 Hz amplitude 1 mm will be selected.
  Arms: Gastrosoleus Muscle Complex Vibration Group
Other: Control Exercise — Lumbar spinal stabilization exerciseswill be given. Lumbar spinal stabilization exercises; Diaphragmatic breathing, and contraction of the transversus abdominis and multifidus muscles will be taught in the supine position. Activation of these muscles will be studied in different positions (prone, crawling, sitting, and sitting on different surfaces). The focus will be on increasing kinesthetic awareness. It will be desirable to ensure and maintain the activation of these muscles during subsequent exercises. Exercises will be continued according to the patient's functional status and individual needs. Advancement of exercises; extremity movements on dynamic surfaces, narrowing of support surfaces, reciprocal movements, increasing the number of resistance and repetitions. The duration of a session will be 40 minutes.
  Arms: Control Exercise Group

SUMMARY:
The aim of this study is to investigate the effects of local vibration application applied to different regions on postural control in addition to spinal stabilization training in ataxic multiple sclerosis (MS) patients.

The study was planned as a single-blind, randomized controlled trial. The patients included in the study will be divided into 3 groups by the closed-envelope randomization method. Each treatment will be 8 weeks, 3 days a week. The control group will be given 40 minutes of lumbar spinal stabilization exercises. Paraspinal vibration group; In addition to 40 minutes of lumbar spinal stabilization exercises, LV will be applied to the paraspinal muscles for 10 minutes. LV application will be applied to the cervical paraspinal muscles for 5 minutes and to the lumbar paraspinal muscles for 5 minutes, bilaterally, sequentially. Gastrosoleus vibration group; In addition to 40 minutes of lumbar spinal stabilization exercises, LV will be applied to the gastrosoleus muscle complex for 10 minutes. LV application will be applied bilaterally, sequentially (5 minutes on the right and left). Assessments will be made by a blind assessor. In assessments; demographic information, Expanded Disability Status Scale (EDSS) /Extended Disability Status Scale (disease stage), International Cooperative Ataxia Rating Scale (ataxia severity), Berg Balance Scale (performance-based balance), Trunk Impairment Scale (trunk control), Neurocom Balance Master Static Posturography (limits of stability and postural sway), OptoGait (gait analysis), lumbopelvic muscle endurance tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-50
* Having been diagnosed with MS by a neurologist
* EDSS score between 3-5
* EDSS pyramidal system score of 3 or less
* Not using corticosteroids and/or stopping at least 3 months before starting the study

Exclusion Criteria:

* Having a history of attacks in the last 3 months
* Having orthopedic or systemic problems
* Presence of peripheral vestibular complaints
* Participating in another exercise program in the last 6 months
* Being mentally affected (Mini-Mental Test Score < 24)
* Severe spasticity (MAS>3)
* Refusal to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale | Assessment will be done before treatment starts ( on average 15 minutes takes).
  Being between Expanded Disability Status Scale 3-5 and having a pyramidal system score below 3 are among the inclusion criteria. At the beginning of the study, all patients will be evaluated for Expanded Disability Status Scale, and patients who do not meet the criteria will not be included in the study.An increase in the score indicates an increase in the severity of the disease.
International Cooperative Ataxia Rating Scale | Change from International Cooperative Ataxia Rating Scale at 8 weeks (each assessment on average 20 minutes takes).
  It will be used to evaluate the severity of ataxia. International Cooperative Ataxia Rating Scale consists of 4 sub-titles: posture and gait disorders, kinetic functions, speech disorders and oculomotor disorders. The score range is in the range of 0-100, with an increase in the score indicating increased disease severity.
Berg Balance Scale | Change from Berg Balance Scale at 8 weeks (each assessment on average 20 minutes takes).
  BBS is a scale that evaluates performance-based balance and scores the performance of 14 different tasks from 0 (not applicable) to 4 (normal performance). In this scale, which is evaluated over 56 points; scores between 0-20 indicate balance disorder, between 21-40 the balance is acceptable, and scores between 41-56 indicate good balance.
Trunk Impairment Scale | Change from Trunk Impairment Scale at 8 weeks (each assessment on average 10 minutes takes).
  The Trunk Impairment Scale, which will be used to evaluate trunk control, has a total of 17 items, of which 3 are static balance, 10 are dynamic balance, and 4 are the coordination ability of the stabilizer muscles. The total score of 0-23 points is recorded. A high score indicates good trunk control.
Limits of Stability and Postural Sways | Change from limits of stability and postural sways at 8 weeks (each assessment on average 15 minutesutes takes).
  It will be evaluated with Neurocom Balance Master Static Posturography. During the test, the patient is asked to stand on the platform without shoes and socks. The upper extremities are asked to be on the side of the trunk without support and to look forward. Limits of stability are evaluated with eyes open on a firm surface. While the feet are on the force platform, the foot contact is maintained and the person is asked to go in 8 directions (forward, right-forward, right, right-back, back, left-back, left, left-forward) without losing balance. The test is finished when all directions are completed. Postural sway is evaluated in 4 situations; eyes open-firm surface, eyes closed-firm surface, eyes open-foam surface, eyes closed-foam surface. The person is asked to be as stable as possible.
Gait Analysis | Change from gait 8 weeks (each assessment on average 5 minutes takes).
  OptoGait Gait Device (Microgate, Bolzano, Italy).Timing, size, and distance are detected and time-distance characteristics are calculated automatically when patients pass between 2 bars positioned on either side of the treadmill. During the test, the patient is asked to get on the treadmill. Then the patient is asked to adjust the speed of the treadmill according to himself (at the speed he feels comfortable) and walk for 1 minute. When the patient walks on the treadmill, objective data about the time-distance characteristics of his gait are obtained. Gait velocity will be recorded in meters/second. Cadence will be recorded in steps/minute.The stride length will be recorded in centimeters.The stance phase and swing phase will be recorded in percent (%).
Prone Bridge Test | Change from lumbopelvic muscle endurance at 8 weeks . In the test, how many seconds they stop is tested.
  Test will be used to evaluate the endurance of lumbopelvic muscles.The patients placed elbows and forearms below their shoulders, straightened the legs. Next, they kept their forearms and toes on the floor, lifted hips, and maintained this straight position as long as possible.
Lateral Bridge Test | Change from lumbopelvic muscle endurance at 8 weeks . In the test, how many seconds they stop is tested.
  Test will be used to evaluate the endurance of lumbopelvic muscles. The patients lay on their left / right sides with support from the forearm with elbows below the shoulders and extended their legs straight. Then the patients lifted their hip from the floor. The test was terminated when the side bridge position deteriorated or the hip fell.
Sorensen Test (Trunk Extensor Test) | Change from lumbopelvic muscle endurance at 8 weeks . In the test, how many seconds they stop is tested.
  Test will be used to evaluate the endurance of lumbopelvic muscles. The patients lied down on a treatment table, aligning their anterior superior iliac spine with the edge of the table, which allowed the upper body to be planked out over the edge. An assessor fixed the patients' pelvis, hip, and knees to the treatment table. The body and the upper extremities were supported using a chair. Next, the chair was removed, and the patients maintained the horizontal body position as long as possible with their arms crossed position on the chest.
Trunk Flexors Test | Change from lumbopelvic muscle endurance at 8 weeks . In the test, how many seconds they stop is tested.
  Test will be used to evaluate the endurance of lumbopelvic muscles. The patients were in a sit-up position while their trunks were supported at the angle of 60 degrees from the floor. They flexed knees and hips at 90 degrees and crossed arms over the chest. Then, the support of the trunk was removed, and the patients maintained this position as long as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kılınç, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No